CLINICAL TRIAL: NCT01096459
Title: Safety and Efficacy of Nerve Rerouting for Treating Neurogenic Bladder in Spina Bifida
Brief Title: Nerve Rerouting Treatment for Neurogenic Bladder in Spina Bifida
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol as presented by investigator was not approved by the NIDDK.
Sponsor: Kenneth Peters, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Kenneth Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-029; R01DK084034 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-31 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Spina Bifida
Keywords: spina; bifida; restore; urinary; function; nerve; reroute
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Nerve Rerouting — All subjects will receive the unilateral nerve rerouting procedure.

SUMMARY:
The goal of this study is to evaluate a surgical procedure (operation) that reroutes lumbar to sacral nerves in the spinal column to improve the bladder's ability to empty properly in patients born with Spina Bifida.

DETAILED DESCRIPTION:
Spina Bifida (a congenital defect of the spinal cord), causes nerve damage and a loss of sensation and muscle function below the waist resulting in bowel and bladder dysfunction. Patients cannot urinate or are constantly wet, and this continues throughout life causing major quality of life and health problems. Clean intermittent catheterization (draining urine from the bladder with a tube) is usually needed to empty the bladder properly. Medications are routinely required to alleviate high urinary tract pressures that can cause irreversible kidney damage, where dialysis or kidney transplant is the only way to sustain life.

A Chinese urologist developed a novel procedure to connect a functioning, healthy lumbar spinal nerve to the sacral nerve that controls the bladder. Hundreds of these procedures have been done in China. The end result is the creation of a new reflex where the bladder can be emptied by scratching or stimulating the skin (over the hip or thigh) supplied by that spinal nerve root. The Chinese physician had reported that of 92 SCI patients, 88% regained bladder control within one year after the nerve rerouting surgery and in 110 children with spina bifida, the reported success was 87% at one year. However, in China rigorous follow up is challenging, therefore much is still unknown about how the nerves regenerate post surgery, complications and results occurring in the first year in particular, and the potential role that central nervous system remodeling may play in achieving successful outcomes. Beaumont urologists were the first in the US to perform this surgery on children with spina bifida. Our preliminary data are very promising, and in 9 subjects at 12 months post procedure, 7/9 subjects could void either voluntarily or by stimulating the new reflex mechanism.

This current project aims to expand upon our pilot experience to conduct a larger and more rigorous study to establish the safety and effectiveness of the proposed somatic-autonomic reflex pathway procedure in gaining bladder and bowel control in patients with spina bifida. We will also collaborate with and train investigators at another site(s) to determine the training needed to achieve similar safety and effectiveness outcomes, and evaluate possible methods to stimulate the new reflex to improve bladder emptying. Achieving the aims outlined in this multicenter proposal will help firmly establish the procedure as safe and effective, and revolutionize the treatment of bladder and bowel dysfunction in patients with spina bifida in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 5 and older with spinal dysraphism (ie. myelomeningocele , lipomyelomeningocele, myelocele, meningocele, occulta) with voiding dysfunction on a CIC program for bladder management for at least one year prior to screening.
2. Atonic or hyperreflexic bladder documented by urodynamic testing during screening. .
3. Documented history of no more than one tethered cord surgery/release in the past; must be > 2 years post tethered cord surgery/release
4. Stable neurogenic bladder dysfunction of at least 1 year or more
5. Normal renal function (cr<1.5 mg/dl or GFR >75)
6. Ambulate independently with or without ankle-foot orthotics (AFOs).
7. Catheterized volume must be at least 50% of total bladder capacity.

Exclusion Criteria:

1. History of bladder cancer, augmentation, or radiation
2. Anatomic outlet obstruction or urethral strictures
3. History of untreated vesico-ureteric reflux grade 4 or higher documented on screening video UDT
4. Hydronephrosis grade 3 or higher
5. Presence of an ileal conduit or supra-pubic catheter drainage
6. Subjects with an artificial bladder sphincter
7. Subjects who have had a sling procedure
8. Subjects who have had the mitrofanoff procedure
9. Bladder botox injections within last 12 months
10. Spina Bifida subjects who underwent intrauterine closure of their myelomeningocele
11. Unable to ambulate independently with or without AFOs.
12. Subject is pregnant
13. Contraindications to general anesthesia or surgery
14. Inability to complete follow up visits for 2 years
15. Inability to complete (or have parent complete) self administered questionnaires
16. Subject possesses any other characteristics that, per investigator's judgment, deems them unsuitable (eg increases risk, impairs data collection, etc) for the procedure/study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Reproducible bladder contraction | 6 to 24 months post procedure
  The primary aim of this study is reproducible bladder contraction of 15cm/H20 or more with scratching the cutaneous dermatome and no significant contraction with stimulation of the non-operated side.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East